CLINICAL TRIAL: NCT00158275
Title: Integrated Care for Depression and Chronic Back Pain
Brief Title: Combined Interventions for Treating Depression and Chronic Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaiser Permanente (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R34MH070642 (NIH); R34MH070642 (NIH); DSIR 83-ATAS
Record Dates: First submitted 2005-09-07; First posted 2005-09-12 (Estimated); Last update posted 2017-10-13 (Actual); Status verified 2017-10

CONDITIONS: Back Pain; Depression
Keywords: Cognitive behavioral therapy; Problem solving therapy; CBT
MeSH Terms: conditions — Back Pain; Depression | interventions — Cognitive Behavioral Therapy; Antidepressive Agents

ARMS (2):
- Integrated Intervention (Experimental): Participants will receive cognitive behavioral therapy for back pain and antidepressants and/or problem solving therapy for depression. Study visits will initially occur once a week and then taper to once every 2 weeks for the 6-month duration.
  Interventions: Behavioral: Cognitive behavioral therapy; Drug: Antidepressants; Behavioral: Problem solving therapy
- Standard of Care (No Intervention): Participants will receive care as usual from their health care provider.

INTERVENTIONS:
Behavioral: Cognitive behavioral therapy — Cognitive behavioral therapy focuses on identifying and eliminating maladaptive beliefs and thoughts.
  Arms: Integrated Intervention
Drug: Antidepressants — Antidepressant drugs try to eliminate symptoms of depression such as persistent sadness and disinterest in normal or pleasurable activities.
  Arms: Integrated Intervention
Behavioral: Problem solving therapy — Problem solving therapy identifies problems that interfere with everyday functions and that contribute to depression and disability. The treatment then provides compensatory strategies that are designed to bypass the person's cognitive limitations and to improve adaptive functioning in the home environment.
  Arms: Integrated Intervention

SUMMARY:
This study will determine the effectiveness of an intervention consisting of combined strategies in reducing the symptoms of both depression and chronic back pain.

DETAILED DESCRIPTION:
The relationship between depression and back pain is complex. Depression is the most common mental condition associated with chronic back pain. Despite this relationship, many patients with depression and back pain seek treatment only for one of the two conditions, which can worsen the untreated condition. An intervention that reduces the symptoms of both depression and back pain is needed. This study will determine the effectiveness of an integrated intervention in reducing both back pain and depression symptoms.

Participants will be randomly assigned to receive either an integrated intervention or standard of care for 6 months. Participants in the integrated intervention group will receive cognitive behavioral therapy for back pain and antidepressants and/or problem solving therapy for depression. Study visits will initially occur once a week and then taper to once every 2 weeks for the 6-month duration; the time of tapering will depend on participant response to treatment and will be at the investigator's discretion. Depression and back pain symptoms will be assessed in all participants at study entry, at the end of treatment, and 6 months after the end of treatment. The study entry and study completion assessments will occur during study visits. The last assessment will be a telephone interview.

ELIGIBILITY:
Inclusion Criteria:

* Roland back pain score of 7 or greater
* Diagnosis of major depression
* Plan to stay enrolled in Group Health Cooperative for the duration of the study and 1 year after the study

Exclusion Criteria:

* Prior surgery
* Cauda equina syndrome (compression and paralysis of nerve roots)
* Schizophrenia or bipolar disorder treatment within 2 years prior to study entry
* Current or prior psychiatric or psychological care for back pain or depression
* At high risk for suicide

Ages: 25 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2004-10; Primary Completion 2006-08 (Actual); Study Completion 2006-08 (Actual)

PRIMARY OUTCOMES:
Depression patient health questionnaire | Measured at study entry, at the end of treatment, and 6 months after the end of treatment
Back pain limitations | Measured at study entry, at the end of treatment, and 6 months after the end of treatment
Roland disability score | Measured at study entry, at the end of treatment, and 6 months after the end of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Michael R. VonKorff, ScD, Principal Investigator — Kaiser Permanente
Locations (1):
- Group Health Cooperative, Seattle, Washington, United States